CLINICAL TRIAL: NCT02468479
Title: Prognostic Values of Chest/Abdominal Wall Varices and Spider Nevi in Patients
Brief Title: Prognostic Values of Chest/Abdominal Wall Varices and Spider Nevi in Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Doctor, General Hospital of Shenyang Military Region
Other Study IDs: CAWV-LC
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No relevant intervention. — No relevant intervention.

SUMMARY:
Chest/abdominal wall varices and spider nevi are two common presenting signs of liver cirrhosis. Their prognostic values remain unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis.
2. Consecutive admission.
3. Permitted to physical examinations.
4. Informed consents.

Exclusion Criteria:

1. Non-cirrhotic portal hypertension.
2. Malignancy.
3. Uncontrolled infection.
4. Severe chronic diseases.
5. Poor patient compliance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of liver cirrhosis who are consecutively admitted to our department.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Prevalence and type of chest/abdominal wall varices and spider nevi | 1.5 years
  Baseline data
Association between etiology of liver cirrhosis and type of chest/abdominal wall varices and spider nevi | 1.5 years
  Baseline data
Association between degree of liver function and type of chest/abdominal wall varices and spider nevi | 1.5 years
  Baseline data
Effect of chest/abdominal wall varices and spider nevi on survival | 2.5 years or more
  Follow-up data

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Guo, MD, PhD, Principal Investigator — Department of Gastroenterology, General Hospital of Shenyang Military Area
Locations (1):
- Department of Gastroenterology, General Hospital of Shenyang Military Area, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Li H, Wang R, Mendez-Sanchez N, Peng Y, Guo X, Qi X. Impact of spider nevus and subcutaneous collateral vessel of chest/abdominal wall on outcomes of liver cirrhosis. Arch Med Sci. 2019 Mar;15(2):434-448. doi: 10.5114/aoms.2018.74788. Epub 2018 Mar 28. PMID 30899297